CLINICAL TRIAL: NCT05644444
Title: A Two-arm, Parallel-design, Clinical Investigation to Determine the Effectiveness and Safety of a Water-based Personal Lubricant With a Sensory Action and Silicone-based Personal Lubricant With a Sensory Action for the Relief of Intimate Discomfort Associated With Vaginal Dryness
Brief Title: Effectiveness and Safety of a Water-based and a Silicone-based Personal Lubricants With Sensory Action
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reckitt Benckiser Healthcare (UK) Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5025003
Record Dates: First submitted 2022-10-20; First posted 2022-12-09 (Actual); Results first posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-08

CONDITIONS: Dyspareunia; Vaginal Dryness
Keywords: Vaginal lubricant
MeSH Terms: conditions — Dyspareunia

STUDY DESIGN:
Intervention Model Description: The personal lubricants will be tested in a 2-arm parallel-design, where subjects will be randomised to an arm/lubricant. Subjects participating in the both the tolerance and treatment phases will be enrolled into an arm for each which includes the same IP/lubricant throughout both phases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lubricant A and Comparator A (Experimental): The comparator will be tested for oral assessment in the tolerance phase only. Tolerance phase includes oral assessment and vaginal assessment. A 7-Day wash-out period followed by 2 visits. Visit 1 will include baseline assessments and application of allocated IP. Visit 2 will consist of clinical assessment. This is conducted on a sub-set of the population enrolled into the arm using the same IP for the treatment phase.
  Treatment phase includes a 4-week run-in period followed by 2 visits. Visit 1 will include baseline assessments and provision of allocated IP. Visit 2 will consist of clinical assessment.
  Interventions: Device: Lubricant A (sensate water-based personal lubricant) and Comparator A (non-sensate water-based lubricant)
- Lubricant B and Comparator B (Experimental): The comparator will be tested for oral assessment in the tolerance phase only. Tolerance phase includes oral assessment and vaginal assessment. A 7-Day wash-out period followed by 2 visits. Visit 1 will include baseline assessments and application of allocated IP. Visit 2 will consist of clinical assessment. This is conducted on a sub-set of the population enrolled into the arm using the same IP for the treatment phase.
  Treatment phase includes a 4-week run-in period followed by 2 visits. Visit 1 will include baseline assessments and provision of allocated IP. Visit 2 will consist of clinical assessment.
  Interventions: Device: Lubricant B (sensate silicone-based personal lubricant) and Comparator B (non-sensate silicone-based personal lubricant)

INTERVENTIONS:
Device: Lubricant A (sensate water-based personal lubricant) and Comparator A (non-sensate water-based lubricant) — In the tolerance phase, a pea-sized lubricant will be considered a single application for oral assessment and approximately 3g of lubricant will be considered a single application for vaginal assessment.
  In the treatment phase, approximately 3g of lubricant will be considered a single application.
  Arms: Lubricant A and Comparator A
Device: Lubricant B (sensate silicone-based personal lubricant) and Comparator B (non-sensate silicone-based personal lubricant) — In the tolerance phase, a pea-sized lubricant will be considered a single application for oral assessment and approximately 3g of lubricant will be considered a single application for vaginal assessment.
  In the treatment phase, approximately 3g of lubricant will be considered a single application.
  Arms: Lubricant B and Comparator B

SUMMARY:
This clinical investigation will look at the effectiveness and safety of two personal lubricants for the relief of intimate discomfort associated with vaginal dryness.

DETAILED DESCRIPTION:
This is an open label, two-arm, parallel-design clinical investigation determining the effectiveness and safety of two personal lubricants. This clinical investigation consists of two phases, a Tolerance Phase and a Treatment Phase, whereby a sub-set of subjects will enter the Tolerance Phase followed by the Treatment Phase. The remaining subjects will enter the Treatment Phase only.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided written informed consent.
2. Subject is aged at least 18 years.
3. Subject in a mutually monogamous heterosexual relationship (≥3 months) who is sexually active, defined as having sexual intercourse at least once a week.
4. Female subject that agrees to have a gynaecological pelvic examination to ensure no significant disease findings and have intact skin and mucous in the test region assessed by the gynaecologist at all the relevant time points.
5. Female subject that agrees to an oral exam by a dermatologist to ensure no significant disease findings and have intact skin and mucous in the test region.
6. Subjects reporting mild to moderate vaginal dryness and dyspareunia during sex (when not using lubricant) in the past 3 months as confirmed on the Verbal Rating Scale (VRS).
7. Pre-menopausal Inclusion Criteria: Female subject of childbearing potential who is willing to use a highly effective method of contraception throughout the clinical investigation.
8. Post-menopausal Inclusion Criteria: Female subject in post-menopausal phase defined as having amenorrhea (absence of menstruation) for at least 12 months.
9. Post-menopausal Inclusion Criteria: Female subject with premature menopause - surgical menopause or physiological menopause within the last 12 months or after having received chemotherapy.

Exclusion Criteria:

1. Subject who has previously experienced an irritant or allergic reaction to any personal lubricant, vaginal moisturiser or female hygiene product or known to have any contact allergen or allergy/hypersensitivity to the test product ingredients.
2. Female subject with history of mucosal intolerance to warming agents.
3. Female subject with continuous or intermittent oral allergy syndrome or burning mouth syndrome of history of thereof.
4. Female subject with urinary, vaginal infection (fungal, bacterial) or sexually transmitted infection which may affect the study outcomes or the safety of the subject.
5. Female subject that has any condition of the oral cavity as determined by the investigator.
6. Male subject has broken skin or wounds in the intimate area.
7. Female subject with a history of skin disorder, which in the opinion of the investigation will affect study outcome.
8. Female subject with autoimmune conditions or any medical conditions which in the opinion of the investigator could compromise the immune function.
9. Female subject who has used any kind of topical histamine and/or topical hormonal based product in the form of an intravaginal cream or moisturiser for local treatment of vaginal dryness in the past 3 months.
10. Female subject using non-medicated, over the counter product, herbal/natural remedies on the vulva, vaginal opening and inside the vagina and is unwilling to stop at least 7 days prior to screening and throughout the duration of clinical investigation.
11. Female subject showing vaginal prolapse and/or other medical conditions that could interfere with the investigation conduct and participation.
12. Female subject who has had surgical cervical excision or vaginal and/or vulvar procedures, including laser and cosmetic procedures to the vulva or vagina in the previous year.
13. Pre-menopausal Exclusion Criteria: Female subject who is pregnant (as confirmed by a positive pregnancy test), breast-feeding or trying to conceive.
14. Post-Menopausal Exclusion Criteria: Female subject that has had previous episodes of vaginal bleeding of unknown origin within the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirstin Deuble-Bente, Medical Doctor, Principal Investigator — proDERM GmbH
Locations (1):
- proDERM GmbH, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No
IPD will be shared as per local regulations.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A single site single country study where recruitment was conducted from February 2023 to March 2023 via advertising at the clinical site.
Pre-assignment Details: Participants meeting inclusion/exclusion criteria were enrolled and either entered the Tolerance Phase or directly into the Treatment Phase.
Groups:
- Lubricant A: The comparator will be tested for oral assessment in the tolerance phase only. Tolerance phase includes oral assessment and vaginal assessment. A 7-Day wash-out period followed by 2 visits. Visit 1 will include baseline assessments and application of allocated IP. Visit 2 will consist of clinical assessment. This is conducted on a sub-set of the population enrolled into the arm using the same IP for the treatment phase.
  Treatment phase includes a 4-week run-in period followed by 2 visits. Visit 1 will include baseline assessments and provision of allocated IP. Visit 2 will consist of clinical assessment.
  Lubricant A (sensate water-based personal lubricant) and Comparator A (non-sensate water-based lubricant): In the tolerance phase, a pea-sized lubricant will be considered a single application for oral assessment and approximately 3g of lubricant will be considered a single application for vaginal assessment.
  In the treatment phase, approximately 3g of lubricant will be considered a single application.
- Lubricant B: The comparator will be tested for oral assessment in the tolerance phase only. Tolerance phase includes oral assessment and vaginal assessment. A 7-Day wash-out period followed by 2 visits. Visit 1 will include baseline assessments and application of allocated IP. Visit 2 will consist of clinical assessment. This is conducted on a sub-set of the population enrolled into the arm using the same IP for the treatment phase.
  Treatment phase includes a 4-week run-in period followed by 2 visits. Visit 1 will include baseline assessments and provision of allocated IP. Visit 2 will consist of clinical assessment.
  Lubricant B (sensate silicone-based personal lubricant) and Comparator B (non-sensate silicone-based personal lubricant): In the tolerance phase, a pea-sized lubricant will be considered a single application for oral assessment and approximately 3g of lubricant will be considered a single application for vaginal assessment.
  In the treatment phase, approximately 3g of lubricant will be considered a single application.
Period: Tolerance Phase
Arm/Group | Lubricant A | Lubricant B
Started | 24 | 20
Completed | 24 | 18
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 2
Period: Treatment Phase
Arm/Group | Lubricant A | Lubricant B
Started | 66 | 66
Completed | 66 | 64
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lubricant A | Lubricant B | Total
Number analyzed (Participants) | 66 | 66 | 132
Age, Customized [Count of Participants; unit: Participants]
  Female 18-65 years | 33 | 33 | 66
  Male at least 18 years | 33 | 33 | 66
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 33 | 33 | 66
  Male | 33 | 33 | 66
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian (Female) | 30 | 29 | 59
  Asian (Female) | 3 | 3 | 6
  Black (Female) | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 66 | 66 | 132

OUTCOME MEASURES:

1. Primary Outcome: Female Sexual Function Index (FSFI) Score Compared to Baseline
Description: The change in FSFI from the baseline event and at 4-weeks post baseline. The FSFI is a 19-item self-report questionnaire to measure sexual functioning in women. The questionnaire assesses six domains of sexual function (sexual desire, sexual arousal, lubrication, orgasm, satisfaction and pain) and provides a total score for sexual function. For individual domain scores, add the scores of the individual questions that comprise the domain and multiply the sum by the domain factor. Add the six domain scores to obtain the total FSFI score. The range of total score is 2.0-36.0. Higher value represents a higher level of sexual function. This measure is the change in total FSFI score between baseline and end of treatment phase (4 weeks).
Time Frame: 4 weeks after baseline
Population: Female participants who were randomized to enter the Treatment Phase of the investigation
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Lubricant A: Sensate water-based personal lubricant
- Lubricant B: Sensate silicone-based personal lubricant
Arm/Group | Lubricant A | Lubricant B
Number analyzed (Participants) | 33 | 32
score on a scale | 4.14 (4.45) | 5.95 (4.07)

2. Secondary Outcome: Change From Baseline in the Female Sexual Function Index (FSFI) Individual Domain Scores
Description: Change from baseline in the FSFI individual domain scores (desire, arousal, lubrication, orgasm, satisfaction and pain) at 4-weeks post baseline For individual FSFI domain scores, add the scores of the individual questions that comprise the domain and multiply the sum by the domain factor. The range of each score is: Desire 1.2-6.0, Arousal 0-6.0, Lubrication 0-6.0, Orgasm 0-6.0, Satisfaction 0.8-6.0 and Pain 0-6.0. Higher value represents a higher level of individual sexual function. This measure is the change in individual FSFI score between baseline and end of treatment phase (4 weeks).
Time Frame: 4 weeks after baseline
Population: Female participants who were randomized to enter the Treatment Phase of the investigation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lubricant A | Lubricant B
Number analyzed (Participants) | 33 | 32
score on a scale
  Domain Desire | 0.27 (0.77) | 0.17 (0.72)
  Domain Arousal | 0.25 (0.83) | 0.62 (0.95)
  Domain Lubrication | 1.00 (1.04) | 1.39 (0.96)
  Domain Orgasm | 0.81 (1.18) | 0.98 (1.21)
  Domain Satisfaction | 0.44 (1.13) | 0.74 (1.46)
  Domain Pain | 1.37 (1.20) | 1.95 (1.24)

3. Secondary Outcome: Subject Perception of the Personal Lubricants Through Subject Perceived Questions
Description: Subjects' perception of each of the two personal lubricants will be determined through Subject Perceived Questions. Participants ranked a statement (strongly agree, agree, neither agree nor disagree, disagree, strongly disagree) that best described the experience. Answering options "agree/strongly agree" were combined to the category 'agreement'.
Time Frame: Initial application (within 24 hours of intercourse) and after 4 weeks
Population: Female participants who were randomized to enter the Treatment Phase of the investigation.
Measure: Count of Participants; unit: Participants
Arm/Group | Lubricant A | Lubricant B
Number analyzed (Participants) | 33 | 32
Participants
  First penetration - Feel smoother (24 hours): Agreement | 32 | 30
  First penetration - Feel smoother (24 hours): Neither agree nor disagree | 1 | 2
  First penetration - Feel smoother (24 hours): Disagree | 0 | 0
  First penetration - Feel smoother (24 hours): Strongly disagree | 0 | 0
  First penetration - Feel smoother (after 4 weeks): Agreement | 31 | 31
  First penetration - Feel smoother (after 4 weeks): Neither agree nor disagree | 2 | 1
  First penetration - Feel smoother (after 4 weeks): Disagree | 0 | 0
  First penetration - Feel smoother (after 4 weeks): Strongly disagree | 0 | 0
  Continuous penetration - feel smoother (24 hours): Agreement | 27 | 31
  Continuous penetration - feel smoother (24 hours): Neither agree nor disagree | 5 | 1
  Continuous penetration - feel smoother (24 hours): Disagree | 1 | 0
  Continuous penetration - feel smoother (24 hours): Strongly disagree | 0 | 0
  Continuous penetration - feel smoother (after 4 weeks): Agreement | 30 | 31
  Continuous penetration - feel smoother (after 4 weeks): Neither agree nor disagree | 1 | 1
  Continuous penetration - feel smoother (after 4 weeks): Disagree | 2 | 0
  Continuous penetration - feel smoother (after 4 weeks): Strongly disagree | 0 | 0
  The lubricant enhances sexual experience (24 hours): Agreement | 16 | 20
  The lubricant enhances sexual experience (24 hours): Neither agree nor disagree | 9 | 8
  The lubricant enhances sexual experience (24 hours): Disagree | 8 | 4
  The lubricant enhances sexual experience (24 hours): Strongly disagree | 0 | 0
  The lubricant enhances sexual experience (after 4 weeks): Agreement | 19 | 20
  The lubricant enhances sexual experience (after 4 weeks): Neither agree nor disagree | 6 | 6
  The lubricant enhances sexual experience (after 4 weeks): Disagree | 6 | 3
  The lubricant enhances sexual experience (after 4 weeks): Strongly disagree | 2 | 3

4. Secondary Outcome: The Evaluation of Product Effectiveness, Tolerability and Usability (Subjective Opinion)
Description: Participants rated their evaluation of Product Effectiveness, Tolerability and Usability after IP use using the following scale: Very Satisfied, Somewhat Satisfied, Neither Satisfied nor Dissatisfied, Somewhat Dissatisfied, Very Dissatisfied.
Time Frame: 4 weeks after baseline
Population: Female participants who were randomized to enter the Treatment Phase of the investigation.
Measure: Count of Participants; unit: Participants
Arm/Group | Lubricant A | Lubricant B
Number analyzed (Participants) | 33 | 32
Participants
  Effectiveness: Very satisfied | 12 | 17
  Effectiveness: Somewhat satisfied | 14 | 11
  Effectiveness: Neither satisfied nor dissatisfied | 5 | 1
  Effectiveness: Somewhat dissatisfied | 2 | 3
  Effectiveness: Very dissatisfied | 0 | 0
  Tolerability: Very satisfied | 14 | 17
  Tolerability: Somewhat satisfied | 13 | 8
  Tolerability: Neither satisfied nor dissatisfied | 2 | 4
  Tolerability: Somewhat dissatisfied | 3 | 1
  Tolerability: Very dissatisfied | 1 | 2
  Usability: Very satisfied | 18 | 14
  Usability: Somewhat satisfied | 10 | 11
  Usability: Neither satisfied nor dissatisfied | 3 | 5
  Usability: Somewhat dissatisfied | 2 | 2
  Usability: Very dissatisfied | 0 | 0

5. Secondary Outcome: The Impression of Change in the Sexual Intimacy (Subjective Opinion)
Description: Subjects' evaluation of improvement in sexual intimacy will be determined through the Patient Global Impression of Change (PGIC) questionnaire which is presented in a form of the visual analogue scale: -3 (much worse), -2, -1, 0 (no change), 1, 2, 3 (much better)
Time Frame: 4 weeks after baseline
Population: Female participants who were randomized to enter the Treatment Phase of the investigation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lubricant A | Lubricant B
Number analyzed (Participants) | 33 | 32
score on a scale | 1.27 (1.04) | 1.34 (1.26)

6. Secondary Outcome: The Assessment of the Vaginal Epithelial Tolerability (VET)
Description: The gynaecologist made an assessment of the VET based on the vaginal dermal tissue for signs and symptoms of erythema, oedema, vulvar membrane dryness, leucorrhoea by using the 5-point scale: 1 (none), 2 (slight), 3 (minimal), 4 (moderate), 5 (severe)
Time Frame: Baseline, 2 and 24 hours post single application
Population: Female participants who were randomized to enter the Tolerance Phase of the investigation.
Measure: Count of Participants; unit: Participants
Arm/Group | Lubricant A | Lubricant B
Number analyzed (Participants) | 12 | 9
Participants
  Baseline: Erythema | 0 | 3
  Baseline: Oedema | 0 | 1
  Baseline: Vulvar membrane | 1 | 1
  Baseline: Leucorrhoea | 0 | 1
  Baseline: No Sign | 11 | 3
  2 hours post application: Erythema | 0 | 1
  2 hours post application: Oedema | 0 | 1
  2 hours post application: Vulvar membrane | 0 | 0
  2 hours post application: Leucorrhoea | 0 | 0
  2 hours post application: No Sign | 12 | 7
  24 hours post application: Erythema | 1 | 0
  24 hours post application: Oedema | 0 | 0
  24 hours post application: Vulvar membrane | 0 | 0
  24 hours post application: Leucorrhoea | 0 | 0
  24 hours post application: No Sign | 11 | 9

7. Secondary Outcome: Tolerability as Assessed by Subject Perceived Questions
Description: Tolerability of the two personal lubricants was determined through Subject Perceived Questions. Participants ranked a statement (strongly agree, agree, neither agree nor disagree, disagree, strongly disagree) that best described the experience. Answering options "agree/strongly agree" were combined to the category 'agreement'.
Time Frame: 24 hours post single application
Population: Female participants who were randomized to enter the Tolerance Phase of the investigation.
Measure: Count of Participants; unit: Participants
Arm/Group | Lubricant A | Lubricant B
Number analyzed (Participants) | 12 | 9
Participants
  Felt gentle on the skin in the vagina: Agreement | 9 | 8
  Felt gentle on the skin in the vagina: Neither agree nor disagree | 1 | 1
  Felt gentle on the skin in the vagina: Disagree | 2 | 0
  Felt gentle on the skin in the vagina: Strongly disagree | 0 | 0
  Felt gentle on the skin of the vulva: Agreement | 9 | 9
  Felt gentle on the skin of the vulva: Neither agree nor disagree | 1 | 0
  Felt gentle on the skin of the vulva: Disagree | 2 | 0
  Felt gentle on the skin of the vulva: Strongly disagree | 0 | 0

8. Secondary Outcome: The Assessment of Overall Tolerance for Each Participant
Description: The gynaecologist and dermatologist made an assessment of tolerance of each subject for each IP based on measured parameters, any clinical signs of irritancy observed and subject's perception of vulvovaginal and oral mucosal tolerance by using the 5-point scale: very good, good, acceptable, poor, very poor.
Time Frame: 24 hours post single application
Population: Female participants who were randomized to enter the Tolerance Phase of the investigation.
Measure: Count of Participants; unit: Participants
Arm/Group | Lubricant A | Lubricant B
Number analyzed (Participants) | 12 | 9
Participants
  Vulvovaginal tolerance: Very Good | 7 | 5
  Vulvovaginal tolerance: Good | 5 | 4
  Vulvovaginal tolerance: Acceptable | 0 | 0
  Vulvovaginal tolerance: Poor | 0 | 0
  Vulvovaginal tolerance: Very Poor | 0 | 0
  Oral mucosal tolerance: Very Good | 11 | 8
  Oral mucosal tolerance: Good | 0 | 0
  Oral mucosal tolerance: Acceptable | 1 | 1
  Oral mucosal tolerance: Poor | 0 | 0
  Oral mucosal tolerance: Very Poor | 0 | 0

9. Secondary Outcome: The Assessment of Oral Mucosal Tolerance
Description: The dermatologist made an assessment of oral mucosal tolerance based on the signs and symptoms of erythema, erosions, oedema and any other signs of clinical irritancy by using the 5-point scale: 1 (none), 2 (slight), 3 (minimal), 4 (moderate), 5 (severe).
Time Frame: Baseline, 30 minutes, 2 hours and 24 hours post application
Population: Female participants who were randomized to enter the Tolerance Phase of the investigation.
Measure: Count of Participants; unit: Participants
Arm/Group | Lubricant A | Lubricant B
Number analyzed (Participants) | 12 | 9
Participants
  Baseline (Erythema, Erosions, Oedema, Any other signs) | 0 | 0
  30 minutes post application (Erythema, Erosions, Oedema, Any other signs) | 0 | 0
  2 hours post application (Erythema, Erosions, Oedema, Any other signs) | 0 | 0
  24 hours post application (Erythema, Erosions, Oedema, Any other signs) | 0 | 0
  No Sign | 12 | 9

10. Secondary Outcome: Overall Proportion of Participants With Adverse Events/Adverse Device Effects (AEs/ADEs)
Description: Overall proportion of participants with Adverse Events/Adverse Device Effects (AEs/ADEs) i.e. the occurrence of one of more AE/ADE per participant.
Time Frame: 10 weeks
Population: Female and male participants who were enrolled to the investigation. For comparators: Female and male participants who were randomized to enter the Tolerance Phase of the investigation.
Measure: Count of Participants; unit: Participants
Groups:
- Comparator A: non-sensate water-based lubricant
- Comparator B: non-sensate silicone-based lubricant
Arm/Group | Lubricant A | Lubricant B | Comparator A | Comparator B
Number analyzed (Participants) | 66 | 66 | 24 | 20
Participants | 10 | 13 | 0 | 0

ADVERSE EVENTS:
Time Frame: 10 weeks
Description: An AE is any untoward medical occurrence, unintended disease or injury or any untoward clinical signs (including an abnormal laboratory finding) in participants, in the context of an investigation, whether or not related to the investigational product. This includes events that are anticipated as well as unanticipated events. This includes events occurring in the context of a clinical investigation related to the investigational device, the comparator or the procedures involved.
Arm/Group | Lubricant A | Lubricant B | Comparator A | Comparator B
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/66 | 0/24 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/66 | 1/66 | 0/24 | 0/20
Other Adverse Events (participants affected / at risk) | 10/66 | 13/66 | 0/24 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lubricant A (N=66) | Lubricant B (N=66) | Comparator A (N=24) | Comparator B (N=20)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shoulder fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lubricant A (N=66) | Lubricant B (N=66) | Comparator A (N=24) | Comparator B (N=20)
- Oral discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (8) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 4 (11) | 2 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intentional device misuse (Injury, poisoning and procedural complications) | 0 (0) | 4 (13) | 0 (0) | 0 (0)
Muscle spasticity (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal discomfort (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the results of the Study, whether in whole or in part, shall be within the sole and absolute discretion of Reckitt, and PI shall not be entitled to publish any of the data or information arising during the Study without the prior written consent of Reckitt.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/44/NCT05644444/Prot_SAP_000.pdf